CLINICAL TRIAL: NCT06418867
Title: The Effect of Mindfulness Intervention Program on Adolescents' Internet Addiction: Quasi-Experimental Study
Brief Title: The Effect of Mindfulness Intervention Program on Adolescents' Internet Addiction
Acronym: Mindfulness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kemal Elyeli (Other)
Responsible Party: Sponsor-Investigator, Kemal Elyeli, Research Asistant, PhD (c), Near East University, Turkey
Organization: Near East University, Turkey (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NearEastU2
Record Dates: First submitted 2024-05-12; First posted 2024-05-17 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Mindfulness; Internet Addiction Disorder; Adolescent Behavior
Keywords: mindfulness; internet addiction disorder; adolescent behavior
MeSH Terms: conditions — Internet Addiction Disorder; Adolescent Behavior | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Mindfulness intervention group
  Interventions: Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Mindfulness — Mindfulness Practice including 6 sessions with 1 hour for each

SUMMARY:
The Internet shows its presence in areas where human beings are actively involved, from education to health, from entertainment to the investment sector. The integration of the Internet into many areas of human life leads to its intensive use. According to the Global Digital Report, the number of individuals with access to the Internet worldwide at the beginning of 2024 is stated as 5.35 billion, and this number constitutes more than 66% of the total world population. One of the pioneering studies on internet addiction was conducted by Young. In this study, five subtypes of internet addiction were identified. These are cyber sex addiction (obsessive use of adult sites such as cyber sex, cyber porn), cyber relationship addiction (excessive involvement in online relationships), net compulsions (online gambling, shopping and trading), information overload (on websites). and constantly surfing databases) and computer addiction (playing computer games). Considering the sub-dimensions of internet addiction, it is seen that it affects many areas of life, from family life to interpersonal relationships, from social life to economic life. Conscious awareness is the awareness of one's internal state and environment. Mindfulness can help people avoid destructive or automatic habits and reactions by learning to observe their thoughts, feelings, and other momentary experiences without judging or reacting. Acting based on awareness is a much different way of life than the autopilot approach in which the individual carries out his daily routines and activities. In studies, mindfulness is examined not only to prevent the recurrence of addiction, but also as a long-term, ongoing health behavior that supports the recovery of addiction. Determining the effect of a mindfulness-based intervention program applied to adolescent nursing students studying at a university on internet addiction and awareness. is intended.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being in the adolescent age group (17-19 years old)
* Studying in Turkish nursing department

Exclusion Criteria:

• Previous participation in a mindfulness intervention program for internet addiction

Ages: 17 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 605 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Internet Addiction Scale | 3 months
  The scale developed by Gunuç consists of 35 items. The scale consists of four sub-dimensions. These dimensions are "Deprivation", "Difficulty in Control", "Impairment in Functionality" and "Social Isolation". The minimum score to be obtained from the scale is 35 and the maximum score is 175. On the scale score, 35-91 points are considered as the non-addicted group, 92-119 as the threshold group, 120-147 as the risk group and 148-175 as the dependent group. The Cronbach alpha (a) internal consistency coefficient of this scale was found to be 0.94. The internal consistency coefficients for the sub-dimensions are; "Deprivation" is 0.89, "Control difficulty" is 0.90, "Impairment in functionality" is 0.92, and "Social Isolation" is 0.90.
Mindful Awareness Scale | 3 months
  The Mindful Awareness Scale was developed by Brown. This scale measures the tendency to be aware of immediate experiences in daily life. It is a one-dimensional scale with 15 items and a 6-point Likert type. As a result of the reliability analysis, the Cronbach's alpha internal consistency coefficient of the scale was calculated as 0.80 and the test-retest correlation was calculated as 0.8. A minimum of 15 and a maximum of 90 points can be obtained from the scale. As the total scale score increases, the level of conscious awareness increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Near East University, Nicosia, Lefkoşa, Cyprus

IPD SHARING:
Plan to Share IPD: No